CLINICAL TRIAL: NCT05086068
Title: Mechanistic and Clinical Study of Intra-articular Arthrosamid for Knee Osteoarthritis
Brief Title: Arthrosamid Injection for OA Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RL1 840
Record Dates: First submitted 2021-10-01; First posted 2021-10-20 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single site, single group of patients identified as requiring treatment for early Osteoarthritis of the knee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arthrosamid Inj (Other): Single arm study - no comparator
  Interventions: Device: Arthrosamid

INTERVENTIONS:
Device: Arthrosamid — Intra-articular hydrogel injection comprising of water and cross-linked polyacrylamide.

SUMMARY:
Prior to surgical intervention, the conservative treatment of knee osteoarthritis involves analgesia and intra-articular injections and currently only steroid injections are available as part of NHS treatment. They have short-term benefit only (<6months) and potentially have detrimental effects on residual cartilage. Arthrosamid is a hydrogel consisting of 97.5% sterile water and 2.5% cross-linked polyacrylamide. It's been shown to be safe and effective, with benefits lasting beyond 2 years in the majority. However, currently it is unclear via what biological pathways it reduces joint inflammation and pain.

This study will investigate the effects of Arthrosamid clinically and biologically.

DETAILED DESCRIPTION:
Prior to surgical intervention, the conservative treatment of knee osteoarthritis involves analgesia and intra-articular injections. Currently only steroid injections are available as part of NHS treatment. It is recognised they have short-term benefit only (<6months) and potentially have detrimental effects on residual cartilage. Arthrosamid is a hydrogel consisting of 97.5% sterile water and 2.5% cross-linked polyacrylamide. It's been shown to be safe and effective, with benefits lasting beyond 2 years in the majority. However, currently it is unclear via what biological pathways it reduces joint inflammation and pain.

Patients with osteoarthritis who are offered an intra-articular knee injection as part of standard care will be asked to enter the trial. On entering the trial baseline outcome measures will be recorded. The level of knee pain will be evaluated using Visual Analogue Scale (VAS). Patients will also be asked to complete the Knee injury and Osteoarthritis Outcome Score (KOOS) score and Western Ontario and McMaster Universities Arthritis Index (WOMAC). Patients will also declare the quantity of anti-inflammatory drugs and Oral analgesia that they have consumed.

At the time of treatment, a blood sample will be taken and under sterile conditions, synovial fluid will be aspirated from the knee prior to 6mls of Arthrosamid being injected. Patients will be reviewed by a researcher in a dedicated research clinic at 3,6 and 12 months post injection and the outcome measures repeated. At 3 months post injection synovial fluid and blood will again be collected from the patients. The blood and synovial fluid pre and post injection in patients who respond well to the injection will be compared to the samples from patients who fail to respond. The differences between the biochemical environments will allow us to identify likely pathways by which the injection reduces pain and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Primary OA according to the American College of Rheumatology criteria1.
* Self-reported pain, aching, or stiffness of the index knee on most days of the past month, and a knee pain score of greater than 40 out of 100 on a visual analogue scale (VAS).
* Radiological OA greater than Kellgren-Lawrence (K-L) grading scale 2
* Patients aged over 18 years
* Patient willing to undergo synovial sampling at 3 months post injection.

Exclusion Criteria:

* Previous trauma with significant alteration in bone architecture
* Symptoms of spinal disease
* Prior injection in the last 12 months
* Joint re-placement operation on the other knee
* Cognitive disorders
* Inflammatory arthritis (i.e., rheumatoid arthritis, spondylarthritis and gout)
* Fibromyalgia
* Auto-immune disease (i.e., connective tissue disorders)
* Previous history of septic arthritis.
* Unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score between baseline (pre-injection) and 6 months and 12 months post-injection. | 6 months and 12 months post injection
  The WOMAC score includes 3 subscales related to pain, stiffness and function; the higher is the WOMAC score, the worse is the joint function.

SECONDARY OUTCOMES:
Blood and synovial fluid biochemical and biomarker levels pre- and post-injection | Pre-injection and at 3 months
  Biochemical and biomarkers to assess clinical effectiveness
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-injection, 3, 6 and 12 months post-injection
  A knee-specific tool, developed to assess the patients' opinion about their knee and associated problems.
Analgesia requirement 1 week prior to Patient Reported Outcome Measurement (PROM) collection | Pre-injection, 3, 6 and 12 months post-injection
  Type and dosage of concomitant medication, specifically analgesia taken in period prior to PROM collection

CONTACTS AND LOCATIONS:
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No